CLINICAL TRIAL: NCT05919693
Title: A 2-part Study Consisting of an Open-label Multiple Ascending Dose (MAD) Safety Study, and a Dose-finding Single-masked Comparative Safety and Preliminary Efficacy Study of Intravitreal (IVT) EYE103 in a Mixed Population of Participants With Diabetic Macular Edema (DME) or Neovascular Age-related Macular Degeneration (NVAMD)
Brief Title: A 2-part Study Consisting of Multiple Ascending Dose (MAD) Safety Study, and a Dose-finding Masked Study to Assess the Safety and Efficacy of Intravitreal (IVT) EYE103 in Patients With Diabetic Macular Edema (DME) or Neovascular Age-related Macular Degeneration (NVAMD)
Acronym: AMARONE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EyeBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EYE103-101; MK-3000-003 (Other: Merck)
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-related Macular Degeneration (NVAMD); Diabetic Macular Edema (DME)
Keywords: Neovascular Age-related Macular Degeneration (NVAMD); Diabetic Macular Edema (DME); Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Part 1 is a multiple-dose escalation study and patients will be enrolled sequentially in ascending order through the dose levels until the highest level is reached or until a maximum tolerated dose is reached, whichever comes first.
  Part 2 is randomized single-masked study where patients on all arms will be enrolled in parallel.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant Care Provider Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose 1 (Experimental): Part 1 MAD Portion Dose 1 - Low Dose
  Interventions: Drug: EYE103
- Dose 2 (Experimental): Part 1 MAD Portion Dose 2 - Low-Mid Dose
  Interventions: Drug: EYE103
- Dose 3 (Experimental): Part 1 MAD Portion Dose 3 - Mid-High Dose
  Interventions: Drug: EYE103
- Dose 4 (Experimental): Part 1 MAD Portion Dose 4 - High Dose
  Interventions: Drug: EYE103
- DME Medium Dose (Experimental): Part 2 Naïve DME monotherapy Medium Dose
  Interventions: Drug: EYE103
- DME High Dose (Experimental): Part 2 Naïve DME monotherapy High Dose
  Interventions: Drug: EYE103
- Naïve NVAMD Medium Dose (Experimental): Part 2 Naïve NVAMD combination therapy Medium Dose
  Interventions: Drug: EYE103
- Naïve NVAMD High Dose (Experimental): Part 2 Naïve NVAMD combination therapy High Dose
  Interventions: Drug: EYE103
- Experienced NVAMD Medium Dose (Experimental): Part 2 Experienced NVAMD combination therapy Medium Dose
  Interventions: Drug: EYE103
- Experienced NVAMD High Dose (Experimental): Part 2 Experienced NVAMD combination therapy High Dose
  Interventions: Drug: EYE103

INTERVENTIONS:
Drug: EYE103 — EYE103 is a humanized antibody formulated for IVT administration

SUMMARY:
EYE103-101 is a 2-part study assessing safety and preliminary efficacy of EYE103 in patients with diabetic macular edema (DME) given as monotherapy or neovascular macular degeneration (NVAMD) given in combination with anti-VEGF.

In the first part, termed the multiple ascending dose (MAD) portion of study, the safety of EYE103 will be assessed at escalating doses. Approximately 12 participants will be entered in this part of the study.

In the second part of the study, called the dose finding part two doses of EYE103 will be selected and their effectiveness will be compared. Approximately 80 participants will be entered in this part of the study.

DETAILED DESCRIPTION:
EYE103-101 is a 2-part study assessing safety and preliminary efficacy of EYE103 in patients with diabetic macular edema (DME) given as monotherapy or neovascular macular degeneration (NVAMD) given in combination with anti-VEGF.

In the first part, termed the multiple ascending dose (MAD) portion of study, the safety of EYE103 will be assessed at escalating doses. Approximately 12 participants will be entered in this part of the study.

In the second part of the study, called the dose finding part two doses of EYE103 will be selected and their effectiveness will be compared. Approximately 80 participants will be entered in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand the study procedures and the risks involved and provide written informed consent before the first study-related activity
* DME patients must be ≥ 18 years of age, NVAMD patients must be ≥ 50 years of age
* Diagnosis of either DME or NVAMD. DME patients must be treatment naïve. NVAMD patients can be either treatment naïve or treatment experienced.
* DME patients must have vision loss in the study eye
* NVAMD patients can be either treatment-naïve or treatment experienced with vision loss in the study eye

Exclusion Criteria:

* Be pregnant or breastfeeding
* History of cataract surgery and/or minimally invasive glaucoma surgery (MIGS) within 3 months of Screening
* Yttrium-Aluminum Garnet (YAG) laser capsulotomy within 2 months of Screening
* Any other condition except for DME or NVAMD or that could affect interpretation of study assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 months
  Adverse Events

SECONDARY OUTCOMES:
Best-corrected Visual Acuity | 3 months
  Best-corrected Visual Acuity

CONTACTS AND LOCATIONS:
Locations (31):
- United States (26):
  - Phoenix, AZ, Phoenix, Arizona
  - Bakersfield, CA, Bakersfield, California
  - Modesto, CA, Modesto, California
  - Mountain View, CA, Mountain View, California
  - Sacramento, CA, Sacramento, California
  - Colorado Springs, Colorado, Colorado Springs, Colorado
  - Lakewood, CO, Lakewood, Colorado
  - Pompano Beach, Pompano Beach, Florida
  - Lemont, NV, Lemont, Illinois
  - Hagerstown, MD, Hagerstown, Maryland
  - Reno, NV, Reno, Nevada
  - West Columbia, SC, West Columbia, South Carolina
  - Germantown, TN, Germantown, Tennessee
  - Knoxville, TN, Knoxville, Tennessee
  - Nashville, TN, Nashville, Tennessee
  - Abilene, TX, Abilene, Texas
  - Amarillo, TX, Amarillo, Texas
  - Austin, TX, Austin, Texas
  - Bellaire, TX, Bellaire, Texas
  - Dallas, TX, Dallas, Texas
  - Katy, TX, Katy, Texas
  - McAllen, TX, McAllen, Texas
  - Plano, TX, Plano, Texas
  - Round Rock, TX, Round Rock, Texas
  - San Antonio, TX, San Antonio, Texas
  - The Woodlands, TX, The Woodlands, Texas
- Argentina (2):
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Caba, Argentina, Caba
- Arecibo, PR, Arecibo, PR, Puerto Rico
- United Kingdom (2):
  - London, England, London, England
  - London, UK, London

IPD SHARING:
Plan to Share IPD: No